CLINICAL TRIAL: NCT02267928
Title: Information Presentation Formats and Pursuit of Diagnostic Information
Brief Title: Information Presentation Formats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Eric VanEpps, PhD Candidate, Carnegie Mellon University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: HS14-574
Record Dates: First submitted 2014-10-14; First posted 2014-10-20 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Meningioma
Keywords: Symptom Assessment
MeSH Terms: conditions — Meningioma | interventions — Coping Orientation to Problems Experienced Questionnaire

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Check/Experience (Experimental): Participants are asked to check the symptoms that they have experienced in the last 6 weeks.
  Interventions: Other: Check Symptoms; Other: Experienced
- Un-check/Experience (Experimental): Participants are asked to un-check the symptoms that they have experienced in the last 6 weeks.
  Interventions: Other: Uncheck Symptoms; Other: Experienced
- Check/Not Experienced (Experimental): Participants are asked to check the symptoms that they have NOT experienced in the last 6 weeks.
  Interventions: Other: Check Symptoms; Other: Not Experienced
- Un-check/Not Experienced (Experimental): Participants are asked to un-check the symptoms that they have NOT experienced in the last 6 weeks.
  Interventions: Other: Uncheck Symptoms; Other: Not Experienced

INTERVENTIONS:
Other: Check Symptoms — Symptoms are "Checked"
  Arms: Check/Experience; Check/Not Experienced
Other: Uncheck Symptoms — Symptoms are "Un-checked"
  Arms: Un-check/Experience; Un-check/Not Experienced
Other: Experienced — Focus of instructions is on symptoms the participant has experienced
  Arms: Check/Experience; Un-check/Experience
Other: Not Experienced — Focus of instructions is on symptoms the participant has NOT experienced
  Arms: Check/Not Experienced; Un-check/Not Experienced

SUMMARY:
Prevention and early detection of medical problems can greatly reduce health care costs, yet time and again, people avoid or ignore services that could help detect medical problems early enough to prevent or reduce the severity of potential problems. The investigators seek to understand whether the elicitation of symptom admission by patients can predict people's perceived risk of the medical condition and voluntary pursuit of medical information.

DETAILED DESCRIPTION:
We will present individuals with medically accurate information about a medical condition and measure people's perceptions of their own likelihood to having that medical condition. This will include an opportunity for people to pursue more information by directing them to a website that features more information about the condition. The initial information provision will vary slightly in presentation (method of eliciting symptoms will vary), and the rate at which individuals visit the subsequent medical website to receive more information will be recorded as a measure of information seeking behavior. Rates will be compared across symptom elicitation conditions to determine which formats are most effective at encouraging information seeking about health issues. No personally identifying information will be collected, and all results will be reported in aggregate. Critically, no deception will be used: Participants will only be provided with information that is as accurate as possible (given existing knowledge in the health/medical fields).

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* American

Exclusion Criteria:

* Mechanical Turk approval rate below 95%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of symptoms | 1 day
  The number of symptoms checked off by participants
Risk of meningioma | 1 day
  Self-reported perceived risk of meningioma
Information pursuit | 1 day
  Binary measure of whether participants click to receive information about meningioma

SECONDARY OUTCOMES:
Funding allocation | 1 day
  Hypothetical federal funding allocation to meningioma
Risk of serious disease | 1 day
  Perceived risk of having any serious disease

CONTACTS AND LOCATIONS:
Overall Officials: Eric M VanEpps, MS, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States